CLINICAL TRIAL: NCT00863772
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED MULTICENTER STUDY OF TANEZUMAB ON PERIPHERAL NERVE FUNCTION IN PATIENTS WITH OSTEOARTHRITIS.
Brief Title: Tanezumab and Nerve Function In Arthritis Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091026; NERVE SAFETY STUDY (Other: Alias Study Number)
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2020-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tanezumab 5 mg (Experimental)
  Interventions: Biological: tanezumab
- Tanezumab 10 mg (Experimental)
  Interventions: Biological: tanezumab
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: tanezumab — 5 mg dose Intravenously every 8 weeks for duration of study
  Arms: Tanezumab 5 mg
Biological: tanezumab — 10 mg dose Intravenously every 8 weeks for duration of study
  Arms: Tanezumab 10 mg
Other: Placebo — Placebo, Intravenously, every 8 weeks for duration of study
  Arms: Placebo

SUMMARY:
Tanezumab reduces pain of osteoarthritis without affecting how nerve impulses are transmitted in sensory nerves.

DETAILED DESCRIPTION:
This study was terminated on 16 Nov 2010 following a US FDA clinical hold for tanezumab osteoarthritis clinical studies which halted dosing and enrollment of patients on 23 June 2010 for potential safety issues.

ELIGIBILITY:
Inclusion Criteria:

* BMI less or equal to 39 kg/m2
* Osteoarthritis (arthritis) of the knee or hip with pain score that qualifies
* Willing to comply with study visit schedule and study requirements, including, for women of child-bearing potential or male patients with female partners of child-bearing potential, the use of 2 forms of birth control, one of which is a barrier method.
* Patients must consent in writing to participate in the study.

Exclusion Criteria:

* Untreated, uncontrolled diseases,
* Unwilling or unable to discontinue the use of prohibited medications, including other pain medications, during the screening period and during the study,
* Significant cardiac disease within the past 6 months
* Significant neurological disease (e.g. peripheral neuropathy, multiple sclerosis, stroke) or signs of neuropathy at screening
* Known bleeding disorder or anticoagulation therapy
* Planned surgery during the study period
* History of alcoholism or drug abuse in the past 2 years
* Unable to use acetaminophen
* Use of a biologic (including live vaccines, with the exception of Flumist) within the past 3 months
* Allergic reaction to a biologic or an antibody in the past
* Disqualifying laboratory values, including Hepatitis B or C, HIV or drug test
* Cancer in the past 5 years. Basal cell or squamous cell carcinoma are okay.
* Medical condition that may interfere with study endpoints or safety of the subject as determined by the investigator.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2009-05-18 (Actual); Primary Completion 2010-11-16 (Actual); Study Completion 2010-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (95):
- United States (95):
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - JDP Medical Research, LLC, Aurora, Colorado
  - Alpine Neurology, Centennial, Colorado
  - Peak Anesthesia, Centennial, Colorado
  - JEM Research, LLC, Atlantis, Florida
  - Medical Specialists of the Palm Beaches, Atlantis, Florida
  - Bradenton Research Center, Inc, Bradenton, Florida
  - Manatee Internal Medicine, Bradenton, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - Harris Bonnette, MD, Fort Myers, Florida
  - Sunrise Clinical Research, Inc., Hollywood, Florida
  - Sunrise Clinical Research, Inc, Hollywood, Florida
  - Pharmax Research Clinic, Inc, Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - Pines Neurological Associates, Pembroke Pines, Florida
  - Pembroke Clinical Trials, Pembroke Pines, Florida
  - Advent Clinical Research Centers, Inc, Pinellas Park, Florida
  - Advent Clinical Research Center, Pinellas Park, Florida
  - Berma Research Group, Plantation, Florida
  - Kennedy-White Orthopaedic Center, Sarasota, Florida
  - Ronal Aung-Din, MD, Sarasota, Florida
  - Ronald Aung-Din, MD, Sarasota, Florida
  - Sarasota Center for Clinical Research, Sarasota, Florida
  - Arthritis & Rheumatic Care Center, South Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - Neuroscience Consultants, LLC, South Miami, Florida
  - Carol L. Pappas MD, PhD, St. Petersburg, Florida
  - Carol L. Pappas, M.D. PhD, St. Petersburg, Florida
  - Dale G. Bramlet, MD, P.L., St. Petersburg, Florida
  - Tampa Neurology Associates, Tampa, Florida
  - Tampa Medical Group, P.A., Tampa, Florida
  - Radiology Associates of Venice & Englewood, Venice, Florida
  - Lovelace Scientific Resources, Inc, Venice, Florida
  - Venice Arthritis Center, Venice, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Atlanta Neurology, Atlanta, Georgia
  - Diagnostic Imaging of Atlanta, Atlanta, Georgia
  - NeuroTrials Research, Incorporated, Atlanta, Georgia
  - Northwest Neurology, P.C., Austell, Georgia
  - Atlanta Knee and Sports Medicine, Decatur, Georgia
  - Joseph D. Weissman, MD, Decatur, Georgia
  - Neurology Specialists of Decatur, Decatur, Georgia
  - Southeastern Center for Clinical Trials, Decatur, Georgia
  - Jefrey D. Lieberman, MD, Decatur, Georgia
  - Northwestern Lake Forest Hospital Diagnostic Imaging Centers, Bannockburn, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Consultants in Neurology, Ltd., Northbrook, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University Hospital, Indianapolis, Indiana
  - Mayo Clinic Rochester, Rochester, Minnesota
  - G. Timothy Kelly, MD, Las Vegas, Nevada
  - Clinical Neurology Specialists, Las Vegas, Nevada
  - Neurological Associates of Long Island, P.C., Lake Success, New York
  - Andrew J. Porges, M.D. PC, Roslyn, New York
  - Asheville Imaging, Asheville, North Carolina
  - Biltmore Medical Associates, Asheville, North Carolina
  - Clinical Study Center of Asheville, LLC, Asheville, North Carolina
  - Asheville Neurology, Asheville, North Carolina
  - Unifour Medical Research Associates, LLC, Hickory, North Carolina
  - Neurology Associates, PA, Hickory, North Carolina
  - Caldwell Memorial Hospital, Lenoir, North Carolina
  - Northstate Clinical Research, Lenoir, North Carolina
  - Ohio Research Center, Toledo, Ohio
  - Bend Memorial Clinic, Bend, Oregon
  - North Star Neurology, Bend, Oregon
  - Altoona Hospital Campus, Altoona, Pennsylvania
  - Blair Neurologic Associates, Altoona, Pennsylvania
  - Blair Medical Associates, Altoona, Pennsylvania
  - Blair Orthopedic Associates, Inc., Altoona, Pennsylvania
  - Bon Secour Campus, Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Coastal Carolina Research Center in Goose Creek, Goose Creek, South Carolina
  - Tidewater Neurology, Goose Creek, South Carolina
  - AAMR Research Clinic, PA, Amarillo, Texas
  - Amarillo Diagnostic Clinic, Amarillo, Texas
  - Radiant Research, Inc., Dallas, Texas
  - Dr. Michael Vengrow, Dallas, Texas
  - Foundation for Southwest Orthopedic Research, Houston, Texas
  - The Neurology Center, Houston, Texas
  - Paragon Research Center, LLC, San Antonio, Texas
  - Baptist M&S Imaging, San Antonio, Texas
  - Sun Research Institute, San Antonio, Texas
  - Christine L. Truitt, MD, San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Neurodiagnostic Laboratories of San Antonio, Inc., San Antonio, Texas
  - Neurodiagnostic Laboratories of San Antonio, Inc, San Antonio, Texas
  - Radiant Research Inc., San Antonio, Texas
  - IntegraTrials, L.L.C, Arlington, Virginia
  - TLC Neurology, P.L.L.C, Arlington, Virginia
  - Virginia Hospital Center, Arlington, Virginia
  - Hypothe Test, LLC, Roanoke, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Evergreen Neurology and Neurodiagnostics, PLLC, Everett, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Brown MT, Cornblath DR, Koltzenburg M, Gorson KC, Hickman A, Pixton GC, Gaitonde P, Viktrup L, West CR. Peripheral Nerve Safety of Nerve Growth Factor Inhibition by Tanezumab: Pooled Analyses of Phase III Clinical Studies in Over 5000 Patients with Osteoarthritis. Clin Drug Investig. 2023 Jul;43(7):551-563. doi: 10.1007/s40261-023-01286-3. Epub 2023 Jul 18. PMID 37460782
- [Derived] Tive L, Bello AE, Radin D, Schnitzer TJ, Nguyen H, Brown MT, West CR. Pooled analysis of tanezumab efficacy and safety with subgroup analyses of phase III clinical trials in patients with osteoarthritis pain of the knee or hip. J Pain Res. 2019 Mar 19;12:975-995. doi: 10.2147/JPR.S191297. eCollection 2019. PMID 30936738
- [Derived] Brown MT, Herrmann DN, Goldstein M, Burr AM, Smith MD, West CR, Verburg KM, Dyck PJ. Nerve safety of tanezumab, a nerve growth factor inhibitor for pain treatment. J Neurol Sci. 2014 Oct 15;345(1-2):139-47. doi: 10.1016/j.jns.2014.07.028. Epub 2014 Jul 18. PMID 25073573
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091026&StudyName=Tanezumab%20and%20Nerve%20Function%20In%20Arthritis%20Patients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who discontinued due to lack of efficacy or completed the treatment in this study, were eligible to enroll in the safety extension study A4091040 (NCT00960804).
Groups:
- Tanezumab 5 mg: Tanezumab (RN624 or PF-04383119) 5 milligram (mg) intravenous infusion over 5 minutes on Day 1, Week 8 and Week 16.
- Tanezumab 10 mg: Tanezumab (RN624 or PF-04383119) 10 mg intravenous infusion over 5 minutes on Day 1, Week 8 and Week 16.
- Placebo: Placebo matched to tanezumab (RN624 or PF-04383119) intravenous infusion over 5 minutes on Day 1, Week 8 and Week 16.
Period: Overall Study
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Started | 74 | 74 | 72
Treated | 73 | 74 | 72
Completed | 6 | 9 | 11
Not Completed | 68 | 65 | 61
Not completed — Adverse Event | 1 | 4 | 0
Not completed — Lack of Efficacy | 4 | 2 | 4
Not completed — Lost to Follow-up | 5 | 1 | 1
Not completed — Protocol Violation | 2 | 0 | 2
Not completed — Withdrawal by Subject | 4 | 7 | 5
Not completed — Study terminated by sponsor | 44 | 45 | 36
Not completed — Entered extension study | 6 | 4 | 9
Not completed — Other | 1 | 2 | 4
Not completed — Randomized but not Treated | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to- treat (ITT) population included all participants who received at least 1 dose of study medication were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo | Total
Number analyzed (Participants) | 73 | 74 | 72 | 219
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 3 | 4 | 11 | 18
  45 to 64 years | 63 | 53 | 50 | 166
  Greater than or equal to (>=) 65 years | 7 | 17 | 11 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 47 | 39 | 130
  Male | 29 | 27 | 33 | 89

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 5 Nerve Conduction Tests-Normal Deviate and Heart Rate Deep Breathing-Normal Deviate (5NC [nd] + HRdb [nd]) Composite Score at Week 24: Intent to Treat (ITT) Analysis Set
Description: 5NC(nd)+HRdb(nd)composite score included 5 Nerve Conduction Studies(NCS)attributes(peroneal motor nerve distal latency [MNDL],peroneal nerve compound muscle action potential[CMAP],peroneal motor nerve conduction velocity[MNCV],tibial MNDL,sural sensory nerve action potential amplitude [SNAP])and HRdb value. Values of attributes scored as percentile(calculated from distribution of normal values corresponding to participant's baseline demographic characteristics),then expressed as normal deviate(nd)score based on standard normal distribution.Score >0=worse response,less than(<)0=better response compared to normal matched population.Score change>0=worsening,<0=improvement compared to baseline.2 neurological visits(NVs) were conducted both at baseline and Week 24. NCS measurements were collected once at each NV.HRdb measurements were collected twice and highest nd score was selected at each NV. Mean of selected measurements at each NV was calculated to obtain Baseline and Week 24 values.
Time Frame: Baseline, Week 24
Population: Intent to treat (ITT) analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo). Missing values were imputed using last observation carried forward (LOCF) method. Here 'number analyzed' signifies participants who were evaluable at specific time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
normal deviate score
  Baseline | 0.61 (2.96) | 1.52 (2.50) | 0.51 (2.71)
  Change at Week 24: number analyzed (Participants) | 58 | 58 | 61
  Change at Week 24 | 0.18 (2.38) | -0.18 (1.73) | -0.15 (2.18)
Statistical Analysis 1: Comparison: Tanezumab 5 mg vs Placebo; Analysis of co-variance (ANCOVA) model was used with treatment as main effect, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.434, ANCOVA; Least squares (LS) mean difference = 0.29, 95% CI 2-sided [-0.44 to 1.01], Standard Error of Mean 0.37
Statistical Analysis 2: Comparison: Tanezumab 10 mg vs Placebo; ANCOVA model was used with treatment as main effect, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.883, ANCOVA; LS mean difference = 0.05, 95% CI 2-sided [-0.68 to 0.79], Standard Error of Mean 0.37

2. Primary Outcome: Change From Baseline in 5 Nerve Conduction Tests-Normal Deviate and Heart Rate Deep Breathing-Normal Deviate (5NC [nd] + HRdb [nd]) Composite Score at Week 24: Per Protocol Analysis Set (PPAS)
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: PPAS included all randomized participants who received at least 1 dose of intravenous study medication and excluded those who violated the exclusion criterion "significant signs of neuropathy at baseline visits". Missing values were imputed using LOCF method. Here 'number analyzed' signifies participants who were evaluable at specific time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 71 | 73 | 71
normal deviate score
  Baseline | 0.45 (2.83) | 1.46 (2.46) | 0.57 (2.69)
  Change at Week 24: number analyzed (Participants) | 56 | 57 | 60
  Change at Week 24 | 0.13 (2.41) | -0.19 (1.74) | -0.11 (2.17)
Statistical Analysis 1: Comparison: Tanezumab 5 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.720, ANCOVA; LS Mean Difference = 0.13, 95% CI 2-sided [-0.59 to 0.86], Standard Error of Mean 0.37
Statistical Analysis 2: Comparison: Tanezumab 10 mg vs Placebo; ANCOVA model was used with treatment as main effect, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.985, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.73 to 0.74], Standard Error of Mean 0.37

3. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score - Lower Limbs [NIS (LL)] at Week 24
Description: NIS-LL: assess muscle weakness, reflexes, sensation; scored separately for left and right limbs. Components of muscle weakness (hip and knee flexion, hip and knee extension, ankle dorsiflexors, ankle plantar flexors, toe extensors, toe flexors) scored on scale 0 (normal) to 4 (paralysis), higher score=greater weakness. Components of reflexes (quadriceps femoris, triceps surae); sensation (touch pressure, pin-prick, vibration, joint position) scored 0 = normal, 1 = decreased, or 2 = absent. NIS-LL score: sum of scores of NIS items 17-24, 28-29 and 34-37. Total possible NIS-LL score range 0-88, high score = more impairment.
Time Frame: Baseline, Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo). Missing values were imputed using LOCF method. Here 'number analyzed' signifies participants who were evaluable at specific time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
units on a scale
  Baseline | 0.00 (0.00) | 0.08 (0.70) | 0.00 (0.00)
  Change at Week 24: number analyzed (Participants) | 68 | 67 | 70
  Change at Week 24 | 0.21 (0.92) | 0.03 (0.95) | 0.06 (0.38)

4. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 24
Description: NIS: 74 items, assess muscle weakness, reflexes and sensation; scored separately for left, right limbs (37 items for each side). Components of muscle weakness are 24 items and scored on scale 0 (normal) to 4 (paralysis), higher score=greater weakness. Components of reflexes and sensation are 13 items and scored 0 = normal, 1= decreased, or 2 = absent. Total possible NIS score range 0 to 244, higher score = greater impairment.
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
units on a scale
  Baseline | 0.00 (0.00) | 0.09 (0.81) | 0.00 (0.00)
  Change at Week 24: number analyzed (Participants) | 68 | 67 | 70
  Change at Week 24 | 0.26 (1.33) | 0.07 (1.35) | 0.06 (0.38)

5. Secondary Outcome: Change From Baseline in Neuropathy Symptoms and Change (NSC) Score at Week 24
Description: NSC score is the number of the 38 symptom questions where the participants indicated experiencing the symptom to any severity. Total score range: 0 to 38 where higher score indicated more symptoms. A change from Baseline > 0 indicated some symptoms of peripheral neuropathy.
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
units on a scale
  Baseline | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Change at Week 24: number analyzed (Participants) | 68 | 67 | 70
  Change at Week 24 | 0.31 (1.03) | 0.13 (0.57) | 0.11 (0.55)

6. Secondary Outcome: Change From Baseline in Peroneal Compound Muscle Action Potential Amplitude (CMAP) Score at Week 24: ITT Analysis Set
Description: Peroneal motor nerve compound muscle action potential amplitude (in millivolts) was measured using electromyography of the left lower limb. Values were scored as percentiles (calculated from distribution of normal values corresponding to participant's baseline demographic characteristics), then expressed as normal deviate (nd) score based on standard normal distribution. Score <0 indicated worse response and >0 indicated better response than the normal matched population. Score change <0 indicated worsening and >0 indicated improvement as compared to baseline. 2 neurological visits (NVs) were conducted both at baseline and Week 24. Mean of the two NV measurements was calculated to obtain Baseline and Week 24 values.
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
normal deviate score
  Baseline | -0.37 (0.94) | -0.55 (0.85) | -0.09 (0.92)
  Change at Week 24: number analyzed (Participants) | 55 | 58 | 61
  Change at Week 24 | -0.12 (0.65) | -0.11 (0.50) | -0.05 (0.59)

7. Secondary Outcome: Change From Baseline in Peroneal Compound Muscle Action Potential Amplitude (CMAP) Score at Week 24: PPAS
Description: Peroneal motor nerve compound muscle action potential amplitude (in millivolts) was measured using electromyography of the left lower limb. Values were scored as percentiles (calculated from distribution of normal values corresponding to participant's baseline demographic characteristics), then expressed as normal deviate (nd) score based on standard normal distribution. Score <0 indicated worse response and >0 indicated better response than the normal matched population. Score change <0 indicated worsening and >0 indicated improvement as compared to baseline. 2 neurological visits (NVs) were conducted both at baseline and Week 24. Mean of the 2 NV measurements was calculated to obtain Baseline and Week 24 values.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 71 | 73 | 71
normal deviate score
  Baseline | -0.35 (0.94) | -0.55 (0.86) | -0.07 (0.91)
  Change at Week 24: number analyzed (Participants) | 53 | 57 | 60
  Change at Week 24 | -0.10 (0.66) | -0.10 (0.50) | -0.06 (0.59)

8. Secondary Outcome: Change From Baseline in Peroneal Motor Nerve Conduction Velocity (MNCV) Score at Week 24: ITT Analysis Set
Description: Peroneal motor nerve conduction velocity (in meters/second) was measured using electromyography of the left lower limb. Values were scored as percentiles (calculated from distribution of normal values corresponding to participant's baseline demographic characteristics), then expressed as normal deviate (nd) score based on standard normal distribution. Score <0 indicated worse response and >0 indicated better response than the normal matched population. Score change <0 indicated worsening and >0 indicated improvement as compared to baseline. 2 neurological visits (NVs) were conducted both at baseline and Week 24. Mean of the 2 NV measurements was calculated to obtain Baseline and Week 24 values.
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
normal deviate score
  Baseline | 0.75 (1.50) | 0.22 (1.28) | 0.26 (1.52)
  Change at Week 24: number analyzed (Participants) | 55 | 58 | 61
  Change at Week 24 | -0.01 (0.91) | 0.12 (1.03) | -0.04 (0.67)

9. Secondary Outcome: Change From Baseline in Peroneal Motor Nerve Conduction Velocity (MNCV) Score at Week 24: PPAS
Description: as for outcome 8
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 71 | 73 | 71
normal deviate score
  Baseline | 0.76 (1.52) | 0.24 (1.28) | 0.21 (1.48)
  Change at Week 24: number analyzed (Participants) | 53 | 57 | 60
  Change at Week 24 | -0.01 (0.91) | 0.11 (1.04) | -0.04 (0.68)

10. Secondary Outcome: Change From Baseline in Peroneal Motor Nerve Distal Latency (MNDL) Score at Week 24: ITT Analysis Set
Description: Peroneal motor nerve distal latency (in milliseconds) was measured using electromyography of the left lower limb. Values were scored as percentiles (calculated from distribution of normal values corresponding to participant's baseline demographic characteristics), then expressed as normal deviate (nd) score based on standard normal distribution. Score >0 indicated worse response and <0 indicated better response as compared to normal matched population. Score change >0 indicated worsening and <0 indicated improvement as compared to baseline. 2 neurological visits (NVs) were conducted both at baseline and Week 24. Mean of the 2 NV measurements was calculated to obtain Baseline and Week 24 values.
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
normal deviate score
  Baseline | -0.19 (1.27) | 0.01 (1.16) | -0.35 (1.07)
  Change at Week 24: number analyzed (Participants) | 55 | 58 | 61
  Change at Week 24 | -0.03 (0.99) | -0.13 (0.56) | -0.08 (0.77)

11. Secondary Outcome: Change From Baseline in Peroneal Motor Nerve Distal Latency (MNDL) Score at Week 24: PPAS
Description: as for outcome 10
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 71 | 73 | 71
normal deviate score
  Baseline | -0.24 (1.25) | -0.01 (1.15) | -0.32 (1.05)
  Change at Week 24: number analyzed (Participants) | 53 | 57 | 60
  Change at Week 24 | -0.03 (1.01) | -0.14 (0.57) | -0.07 (0.77)

12. Secondary Outcome: Change From Baseline in Tibial Motor Nerve Distal Latency (MNDL) Score at Week 24: ITT Analysis Set
Description: Tibial motor nerve distal latency (in milliseconds) was measured using electromyography of the left lower limb. Values were scored as percentiles (calculated from distribution of normal values corresponding to participant's baseline demographic characteristics), then expressed as normal deviate (nd) score based on standard normal distribution. Score >0 indicated worse response and <0 indicated better response as compared to normal matched population. Score change >0 indicated worsening and <0 indicated improvement as compared to baseline. 2 neurological visits (NVs) were conducted both at baseline and Week 24. Mean of the 2 NV measurements was calculated to obtain Baseline and Week 24 values.
Time Frame: Baseline, Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo). Missing values were imputed using LOCF method. Here 'number analyzed' participants who were evaluable at specific time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
normal deviate score
  Baseline | 0.73 (1.25) | 0.90 (1.18) | 0.83 (1.09)
  Change at Week 24: number analyzed (Participants) | 55 | 58 | 61
  Change at Week 24 | 0.20 (1.08) | -0.16 (0.81) | -0.08 (0.91)

13. Secondary Outcome: Change From Baseline in Tibial Motor Nerve Distal Latency (MNDL) Score at Week 24: PPAS
Description: as for outcome 12
Time Frame: Baseline, Week 24
Population: PPAS included all randomized participants who received at least 1 dose of intravenous study medication and excluded those who violated the exclusion criterion "significant signs of neuropathy at baseline visits". Missing values were imputed using LOCF method. Here, 'number analyzed' signifies participants who were evaluable at specific time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 71 | 73 | 71
normal deviate score
  Baseline | 0.69 (1.24) | 0.90 (1.19) | 0.82 (1.09)
  Change at Week 24: number analyzed (Participants) | 53 | 57 | 60
  Change at Week 24 | 0.20 (1.10) | -0.17 (0.80) | -0.09 (0.92)

14. Secondary Outcome: Change From Baseline in Sural Sensory Nerve Action Potential Amplitude (SNAP) Score at Week 24: ITT Analysis Set
Description: Sural sensory nerve action potential amplitude (in microvolts) was measured using electromyography of the left lower limb. Values were scored as percentiles (calculated from distribution of normal values corresponding to participant's baseline demographic characteristics), then expressed as normal deviate (nd) score based on standard normal distribution. A score <0 indicated worse response and >0 indicated better response than the normal matched population. A change <0 indicated worsening and >0 indicated improvement compared to baseline. 2 neurological visits (NVs) were conducted both at baseline and Week 24. Mean of the 2 NV measurements was calculated to obtain Baseline and Week 24 values.
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
normal deviate score
  Baseline | -0.20 (1.12) | -0.06 (1.00) | -0.22 (1.07)
  Change at Week 24: number analyzed (Participants) | 55 | 58 | 61
  Change at Week 24 | -0.03 (0.97) | -0.12 (0.71) | 0.01 (0.86)

15. Secondary Outcome: Change From Baseline in Sural Sensory Nerve Action Potential Amplitude (SNAP) Score at Week 24: PPAS
Description: as for outcome 14
Time Frame: Baseline, Week 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 71 | 73 | 71
normal deviate score
  Baseline | -0.17 (1.09) | -0.05 (1.00) | -0.25 (1.05)
  Change at Week 24: number analyzed (Participants) | 53 | 57 | 60
  Change at Week 24 | 0.01 (0.93) | -0.12 (0.72) | 0.03 (0.85)

16. Secondary Outcome: Change From Baseline in Heart Rate Deep Breathing [HRdb] at Week 24: ITT Analysis Set
Description: HRdb test was used to evaluate the effect of treatment on autonomic function. Participants took a series of 8 deep breaths and average heart rate difference was measured and compared to normative data. R-R (time between two consecutive R waves in the electrocardiogram) response to deep breathing was reported as a normal deviates. Score <0 indicated worse response and >0 indicated better response as compared to normal matched population. Score change <0 indicated worsening and >0 indicated improvement as compared to baseline. 2 neurological visits (NVs) were conducted both at baseline and Week 24. Measurements of HRdb were collected twice and highest nd score was selected at each NV. Mean of the 2 selected NV measurements was calculated to obtain Baseline and Week 24 values.
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
normal deviate score
  Baseline | -0.25 (0.76) | -0.23 (0.79) | 0.01 (1.05)
  Change at Week 24: number analyzed (Participants) | 56 | 56 | 60
  Change at Week 24 | 0.06 (0.57) | -0.01 (0.66) | 0.02 (0.64)

17. Secondary Outcome: Change From Baseline in Heart Rate Deep Breathing [HRdb] at Week 24: PPAS
Description: as for outcome 16
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 71 | 73 | 71
normal deviate score
  Baseline | -0.23 (0.76) | -0.22 (0.79) | 0.04 (1.04)
  Change at Week 24: number analyzed (Participants) | 54 | 55 | 60
  Change at Week 24 | 0.05 (0.57) | -0.02 (0.66) | 0.02 (0.64)

18. Secondary Outcome: Change From Baseline in 5 Nerve Conduction Test - Normal Deviate [5NC (nd)] at Week 24: ITT Analysis Set
Description: 5NC (nd) score included 5 NCS attributes: peroneal MNDL, CMAP, MNCV, tibial MNDL and sural SNAP. Values of attributes scored as percentiles (calculated from distribution of normal values corresponding to participant's baseline demographic characteristics), then expressed as normal deviate (nd) score based on standard normal distribution. Total score calculated as sum of each NCS attribute. Total score >0 indicated worse and <0 indicated better response as compared to normal matched population. Total score change >0 indicated worsening and <0 indicated improvement as compared to baseline. 2 neurological visits (NVs) were conducted both at baseline and Week 24. Mean of the 2 NV measurements was calculated to obtain Baseline and Week 24 values.
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
normal deviate score
  Baseline | 0.36 (2.86) | 1.30 (2.18) | 0.53 (2.62)
  Change at Week 24: number analyzed (Participants) | 55 | 58 | 61
  Change at Week 24 | 0.34 (2.04) | -0.18 (1.60) | -0.09 (2.03)

19. Secondary Outcome: Change From Baseline in 5 Nerve Conduction Test - Normal Deviate (5NC [nd]) at Week 24: PPAS
Description: 5NC (nd) score included 5 NCS attributes: peroneal MNDL, CMAP, MNCV, tibial MNDL and sural SNAP. Values of attributes scored as percentiles (calculated from distribution of normal values corresponding to participant's baseline demographic characteristics), then expressed as normal deviate (nd) score based on standard normal distribution. Total score calculated as sum of each NCS attribute. Total score >0 indicated worse and <0 indicated better response as compared to normal matched population. Total score change >0 indicated worsening and <0 indicated improvement as compared to baseline.2 neurological visits (NVs) were conducted both at baseline and Week 24. Mean of the 2 NV measurements was calculated to obtain Baseline and Week 24 values.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 71 | 73 | 71
normal deviate score
  Baseline | 0.22 (2.76) | 1.25 (2.15) | 0.60 (2.56)
  Change at Week 24: number analyzed (Participants) | 53 | 57 | 60
  Change at Week 24 | 0.28 (2.05) | -0.20 (1.60) | -0.09 (2.05)

20. Secondary Outcome: Change From Baseline in Protein Gene Product (PGP) 9.5-Positive Intraepidermal Epidermal Nerve Fiber (IENF) Density at Week 24
Description: IENF density was quantified in 3 millimeter (mm) immunostained (PGP 9.5-immunohistochemical staining) skin punch biopsies taken from the distal end of the leg, 10 centimeter (cm) above the lateral malleolus, within the territory of the sural nerve, containing epidermis and superficial dermis to evaluate amount of small diameter nerve fibers. Skin biopsies were taken from normal appearing skin and skin having local scar, signs of trauma, ulceration, or active dermatologic process were avoided.
Time Frame: Baseline, Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo). Missing values imputed using LOCF. Here 'overall number of participants analyzed' signifies participants evaluable for this measure and 'number analyzed' signifies participants evaluable at specific time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: nerve fiber count/millimeter
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 71 | 73 | 71
nerve fiber count/millimeter
  Baseline | 11.61 (6.33) | 11.31 (5.01) | 12.43 (6.48)
  Change at Week 24: number analyzed (Participants) | 52 | 53 | 53
  Change at Week 24 | 0.31 (4.17) | -0.91 (3.86) | -0.52 (4.15)

21. Secondary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Weeks 8, 16, and 24
Description: WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in the index joint (knee or hip) in the past 48 hours. It is calculated as the mean of the scores from the 5 individual questions scored on a numerical rating scale (NRS) of 0 to 10, where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 to 10, where higher scores indicate higher pain.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo). Missing values were imputed using LOCF method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
units on a scale
  Baseline | 5.99 (1.49) | 6.45 (1.34) | 6.54 (1.55)
  Change at Week 8 | -2.09 (2.44) | -2.87 (2.82) | -1.12 (1.78)
  Change at Week 16 | -2.12 (2.22) | -2.56 (2.75) | -1.35 (1.80)
  Change at Week 24 | -2.06 (2.38) | -2.46 (2.68) | -1.39 (1.85)

22. Secondary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Score at Weeks 8, 16, and 24
Description: WOMAC physical function subscale is a 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in the index joint (knee or hip) in the past 48 hours. It is calculated as the mean of the scores from the 17 individual questions scored on a NRS of 0 to 10, where higher scores indicate worse function. Total score range for WOMAC physical function subscale score is 0 to 10, where higher scores indicate worse function.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
units on a scale
  Baseline | 6.04 (1.55) | 6.19 (1.62) | 6.52 (1.70)
  Change at Week 8 | -1.86 (2.44) | -2.90 (2.74) | -1.03 (1.79)
  Change at Week 16 | -1.99 (2.37) | -2.61 (2.68) | -1.15 (1.85)
  Change at Week 24 | -1.97 (2.50) | -2.47 (2.62) | -1.19 (1.82)

23. Secondary Outcome: Change From Baseline in the Patient's Global Assessment (PGA) of Osteoarthritis at Weeks 8, 16, and 24
Description: Participants answered: Considering all the ways your osteoarthritis in your knee or hip affects you, how are you doing today? Participants rated their condition using a 5-point scale where 1 = very good (asymptomatic and no limitation of normal activities), 2 = good (mild symptoms and no limitation of normal activities), 3 = fair (moderate symptoms and limitation of some normal activities), 4 = poor (Severe symptoms and inability to carry out most normal activities) and, 5 =very poor (Very severe symptoms which are intolerable and inability to carry out all normal activities). Higher score indicated severe condition.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
units on a scale
  Baseline | 3.29 (0.51) | 3.28 (0.45) | 3.36 (0.56)
  Change at Week 8 | -0.70 (0.95) | -0.88 (1.08) | -0.46 (0.80)
  Change at Week 16 | -0.78 (0.98) | -0.82 (1.06) | -0.56 (0.82)
  Change at Week 24 | -0.75 (1.00) | -0.74 (1.01) | -0.56 (0.85)

24. Secondary Outcome: Percentage of Participants With Outcome Measures in Rheumatology - Osteoarthritis Research Society International (OMERACT-OARSI) Response
Description: OMERACT-OARSI response: >=50 percent (%) improvement from baseline and absolute change from baseline of >=2 units in WOMAC pain or physical function subscale, or at least 2 of the following 3 being true: >=20% improvement from baseline and absolute change from baseline of >=1 unit in 1) WOMAC pain subscale, 2) WOMAC physical function subscale, 3) PGA of osteoarthritis (score: 1-5, higher score=more affected). WOMAC pain, physical function subscales assess amount of pain/difficulty experienced (score: 0-10, higher score=higher pain/difficulty).
Time Frame: Weeks 8, 16, and 24
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
percentage of participants
  Week 8 | 49.3 | 64.9 | 37.5
  Week 16 | 52.1 | 62.2 | 40.3
  Week 24 | 52.1 | 59.5 | 38.9

25. Secondary Outcome: Percentage of Participants With At Least 30%, 50%, 70% and 90% Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score
Description: The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in the index joint ( knee or hip) in the past 48 hours. It is calculated as the mean of the scores from 5 individual questions scored on a numerical rating scale (NRS) of 0 to 10, where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 to 10, where higher scores indicate higher pain.
Time Frame: Weeks 8, 16, and 24
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
percentage of participants
  Week 8: >=30% Reduction | 46.6 | 56.8 | 30.6
  Week 8: >=50% Reduction | 37.0 | 44.6 | 15.3
  Week 8: >=70% Reduction | 26.0 | 32.4 | 5.6
  Week 8: >=90% Reduction | 15.1 | 18.9 | 2.8
  Week 16: >=30% Reduction | 47.9 | 54.1 | 36.1
  Week 16: >=50% Reduction | 39.7 | 39.2 | 15.3
  Week 16: >=70% Reduction | 24.7 | 27.0 | 9.7
  Week 16: >=90% Reduction | 11.0 | 18.9 | 2.8
  Week 24: >=30% Reduction | 46.6 | 52.7 | 36.1
  Week 24: >=50% Reduction | 35.6 | 37.8 | 20.8
  Week 24: >=70% Reduction | 26.0 | 25.7 | 9.7
  Week 24: >=90% Reduction | 13.7 | 17.6 | 4.2

26. Secondary Outcome: Percentage of Participants With Improvement of At Least 2 Points From Baseline in Patient's Global Assessment (PGA) of Osteoarthritis
Description: as for outcome 23
Time Frame: Weeks 8, 16, and 24
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
percentage of participants
  Week 8 | 19.2 | 31.1 | 8.3
  Week 16 | 21.9 | 29.7 | 12.5
  Week 24 | 21.9 | 27.0 | 9.7

27. Secondary Outcome: Number of Participants With Cumulative Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score
Description: The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in the index joint (knee or hip) in the past 48 hours. It is calculated as the mean of the scores from the 5 individual questions scored on a numerical rating scale (NRS) of 0 to 10, where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 to 10, where higher scores indicate higher pain. Participants with specified reduction (as percent) from baseline at Week 16 are reported.
Time Frame: Week 16
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
Participants
  >0% | 55 | 50 | 51
  >=10% | 45 | 48 | 39
  >=20% | 39 | 46 | 31
  >=30% | 35 | 40 | 26
  >=40% | 34 | 31 | 21
  >=50% | 29 | 29 | 11
  >=60% | 26 | 24 | 9
  >=70% | 18 | 20 | 7
  >=80% | 13 | 15 | 4
  >=90% | 8 | 14 | 2
  100% | 4 | 9 | 0

28. Secondary Outcome: Change From Baseline in Average Pain Score in the Index Knee/Hip Joint at Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15 16, 17, 18, 19, 20, 21, 22, 23, and 24
Description: Participants assessed daily average index joint pain during the past 24 hours on an 11-point NRS ranging from 0 (no pain) to 10 (worst pain). Higher score indicated greater pain.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15 16, 17, 18, 19, 20, 21, 22, 23, and 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
units on a scale
  Baseline | 6.04 (1.73) | 6.33 (1.67) | 6.45 (1.88)
  Change at Week 1 | -1.62 (1.80) | -2.04 (1.97) | -0.75 (1.36)
  Change at Week 2 | -1.88 (2.08) | -2.00 (2.35) | -0.94 (1.81)
  Change at Week 3 | -1.80 (2.26) | -2.13 (2.67) | -0.99 (1.93)
  Change at Week 4 | -2.32 (2.26) | -2.92 (2.79) | -1.05 (1.86)
  Change at Week 5 | -2.46 (2.27) | -2.98 (2.86) | -1.17 (1.87)
  Change at Week 6 | -2.48 (2.31) | -3.00 (2.88) | -1.21 (1.97)
  Change at Week 7 | -2.48 (2.36) | -2.97 (3.04) | -1.21 (1.93)
  Change at Week 8 | -2.46 (2.37) | -2.82 (2.97) | -1.10 (1.81)
  Change at Week 9 | -2.44 (2.41) | -2.87 (2.93) | -1.12 (1.90)
  Change at Week 10 | -2.42 (2.36) | -2.77 (2.85) | -1.32 (2.14)
  Change at Week 11 | -2.33 (2.20) | -2.62 (2.88) | -1.36 (2.12)
  Change at Week 12 | -2.37 (2.28) | -2.72 (2.87) | -1.32 (2.07)
  Change at Week 13 | -2.26 (2.26) | -2.81 (2.94) | -1.26 (2.04)
  Change at Week 14 | -2.35 (2.27) | -2.71 (2.94) | -1.23 (1.88)
  Change at Week 15 | -2.30 (2.23) | -2.74 (2.91) | -1.19 (1.89)
  Change at Week 16 | -2.27 (2.20) | -2.62 (2.88) | -1.15 (1.96)
  Change at Week 17 | -2.33 (2.16) | -2.68 (2.96) | -1.25 (2.07)
  Change at Week 18 | -2.40 (2.33) | -2.71 (2.95) | -1.20 (2.04)
  Change at Week 19 | -2.26 (2.18) | -2.73 (2.90) | -1.17 (1.95)
  Change at Week 20 | -2.32 (2.26) | -2.71 (2.89) | -1.20 (1.88)
  Change at Week 21 | -2.32 (2.24) | -2.74 (2.91) | -1.24 (1.93)
  Change at Week 22 | -2.30 (2.18) | -2.71 (2.89) | -1.29 (2.00)
  Change at Week 23 | -2.30 (2.25) | -2.66 (2.90) | -1.28 (1.97)
  Change at Week 24 | -2.28 (2.30) | -2.64 (2.90) | -1.20 (1.87)

29. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score at Weeks 8, 16, and 24
Description: The WOMAC stiffness subscale is a 2-item questionnaire used to assess the amount of stiffness experienced due to osteoarthritis in the index joint (knee or hip) in the past 48 hours. It is calculated as the mean of the scores from the 2 individual questions scored on NRS of 0 to 10, with higher scores indicating more stiffness. Total score range for WOMAC stiffness subscale score is 0 to 10, where higher scores indicate more stiffness. Stiffness was defined as a sensation of decreased ease of movement in the index joint (knee or hip).
Time Frame: Baseline, Weeks 8, 16, and 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
units on a scale
  Baseline | 6.38 (1.80) | 6.74 (1.62) | 6.72 (1.82)
  Change at Week 8 | -2.14 (2.64) | -3.18 (2.95) | -1.08 (1.92)
  Change at Week 16 | -2.36 (2.53) | -2.84 (2.90) | -1.22 (1.91)
  Change at Week 24 | -2.37 (2.66) | -2.70 (2.86) | -1.33 (2.02)

30. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Weeks 8, 16, and 24
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain (5 items), stiffness (2 items) and physical function (17 items) in participants with osteoarthritis of knee or hip. WOMAC average score is the mean of WOMAC Pain, Physical Function and Stiffness subscale scores and ranges from 0 to 10, where higher score indicates worse response. Change from baseline <0 indicates an improvement.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
units on a scale
  Baseline | 6.14 (1.51) | 6.46 (1.40) | 6.59 (1.62)
  Change at Week 8 | -2.03 (2.41) | -2.98 (2.78) | -1.08 (1.73)
  Change at Week 16 | -2.16 (2.29) | -2.67 (2.71) | -1.24 (1.75)
  Change at Week 24 | -2.13 (2.44) | -2.54 (2.66) | -1.30 (1.80)

31. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale Item: Pain When Walking on a Flat Surface at Weeks 8, 16, and 24
Description: Participants answered: "How much pain have you had when walking on a flat surface?". Participants responded by using a NRS of 0 to 10, where 0 = no pain and 10 = extreme pain. Higher score indicated greater pain. Change from baseline <0 indicated an improvement.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
units on a scale
  Baseline | 5.88 (1.55) | 6.20 (1.52) | 6.47 (1.64)
  Change at Week 8 | -2.01 (2.51) | -2.74 (2.94) | -1.21 (1.96)
  Change at Week 16 | -2.04 (2.26) | -2.53 (2.84) | -1.44 (1.98)
  Change at Week 24 | -1.97 (2.41) | -2.35 (2.75) | -1.38 (1.95)

32. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale Item: Pain When Going Up or Down Stairs at Weeks 8, 16, and 24
Description: Participants answered: How much pain have you had when going up or down stairs?. Participants responded by using a NRS of 0 to 10, where 0 = no pain and 10 = extreme pain. Higher score indicated greater pain. Change from baseline <0 indicates an improvement.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
units on a scale
  Baseline | 7.16 (1.72) | 7.49 (1.30) | 7.61 (1.60)
  Change at Week 8 | -2.30 (2.71) | -3.04 (2.98) | -1.17 (2.05)
  Change at Week 16 | -2.32 (2.49) | -2.74 (2.94) | -1.21 (2.24)
  Change at Week 24 | -2.22 (2.67) | -2.64 (2.87) | -1.18 (2.16)

33. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Domain Scores at Week 24
Description: SF-36v2 is a self-administered questionnaire evaluating 8 aspects/domains of functional health and wellbeing: physical function, role physical, bodily pain, vitality, general health, social function, role emotional and mental health. The total score for each domain is scaled 0-100 (100 = highest level of functioning). Change from baseline >0 indicates an improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
units on a scale
  Baseline: General Health | 72.22 (14.75) | 72.36 (16.39) | 70.85 (20.25)
  Baseline: Physical Function | 38.00 (19.58) | 38.58 (18.50) | 40.28 (23.19)
  Baseline: Role Physical | 53.08 (24.81) | 49.75 (26.26) | 49.57 (27.36)
  Baseline: Bodily Pain | 39.44 (15.53) | 36.36 (14.78) | 37.97 (16.49)
  Baseline: Vitality | 55.74 (19.09) | 56.53 (19.50) | 57.90 (22.15)
  Baseline: Social Function | 72.09 (22.68) | 75.00 (22.38) | 73.96 (25.76)
  Baseline: Role Emotional | 75.23 (26.89) | 74.44 (27.97) | 71.64 (27.71)
  Baseline: Mental Health | 76.78 (16.92) | 77.70 (16.90) | 76.88 (18.30)
  Change at Week 24: General Health | 0.44 (8.57) | 0.72 (5.56) | -0.28 (7.84)
  Change at Week 24: Physical Function | 3.72 (12.34) | 4.66 (12.34) | 3.13 (16.43)
  Change at Week 24: Role Physical | 1.71 (11.47) | 5.74 (15.92) | 5.82 (12.60)
  Change at Week 24: Bodily Pain | 3.25 (13.98) | 6.30 (16.98) | 4.07 (10.88)
  Change at Week 24: Vitality | 1.20 (8.82) | 2.03 (9.82) | 0.52 (6.00)
  Change at Week 24: Social Function | 0.51 (8.70) | 1.86 (15.98) | 0.17 (10.38)
  Change at Week 24: Role Emotional | -2.05 (13.59) | 2.14 (16.09) | 3.70 (15.57)
  Change at Week 24: Mental Health | 0.07 (7.61) | 0.95 (10.19) | -0.42 (5.98)

34. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Physical and Mental Component Scores at Week 24
Description: SF-36v2 is a self-administered questionnaire evaluating 8 aspects/domains of functional health and wellbeing: physical function, role physical, bodily pain, vitality, general health, social function, role emotional and mental health. Total score for each aspect were scaled 0-100(100=highest level of functioning). For obtaining physical and mental component scores, z-score for each scale=(observed score - mean score for general 1990 United States [US] population)/corresponding standard deviation. The 2 component scores were obtained by multiplying each aspect z-score by physical or mental factor score coefficient (1990 general US population) and summing the eight products. Component scores indicated how many standard deviations higher (in case of positive z-score [better functioning])/lower (in case of negative z-score [worse functioning]) participant's value was relative to the mean of the reference population. Change from baseline >0 indicates an improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
Z-score
  Baseline: Mental Component Score | 0.34 (1.09) | 0.42 (1.12) | 0.32 (1.18)
  Baseline: Physical Component Score | -1.54 (0.74) | -1.62 (0.74) | -1.55 (0.82)
  Change at Week 24: Mental Component Score | -0.08 (0.48) | 0.02 (0.57) | -0.00 (0.44)
  Change at Week 24: Physical Component Score | 0.16 (0.52) | 0.23 (0.55) | 0.16 (0.49)

35. Secondary Outcome: Number of Participants With Rescue Medication Usage
Description: In case of inadequate pain relief for osteoarthritis during the treatment period, acetaminophen up to 3000 mg per day up to 3 days per week could be taken as rescue medication.
Time Frame: Week 8, 16, 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo). Missing values were imputed using LOCF method. Here 'overall number of participants analyzed' signifies those participants who were evaluable for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 70 | 71 | 72
Participants
  Week 8 | 25 | 38 | 40
  Week 16 | 23 | 28 | 41
  Week 24 | 23 | 23 | 36

36. Secondary Outcome: Number of Days With Rescue Medication Usage
Description: In case of inadequate pain relief for osteoarthritis during the treatment period, acetaminophen up to 3000 mg per day up to 3 days per week could be taken as rescue medication. Result reported is number of days of rescue medication use in each week, and ranges from 0 to 7.
Time Frame: Weeks 8, 16, and 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo). Missing values were imputed using LOCF method. Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 70 | 71 | 72
days per week
  Week 8 | 1.0 (1.79) | 1.2 (1.64) | 1.4 (1.80)
  Week 16 | 0.9 (1.69) | 0.8 (1.41) | 1.3 (1.80)
  Week 24 | 1.0 (1.85) | 0.7 (1.40) | 1.4 (1.98)

37. Secondary Outcome: Amount of Rescue Medication Used
Description: In case of inadequate pain relief for osteoarthritis during the treatment period, acetaminophen up to 3000 mg per day up to 3 days per week could be taken as rescue medication. Results reported is total dose of acetaminophen (in mg) for each week.
Time Frame: Weeks 8, 16, and 24
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mg per week
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 70 | 71 | 72
mg per week
  Week 8 | 1192.9 (2317.7) | 1422.5 (2391.4) | 2402.8 (3899.8)
  Week 16 | 1128.6 (2270.9) | 1028.2 (2253.4) | 2222.2 (3608.4)
  Week 24 | 1228.6 (2422.2) | 908.5 (2252.5) | 2194.4 (3598.3)

38. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA)
Description: Human serum samples were analyzed for the presence or absence of anti-tanezumab antibodies by using the semiquantitative enzyme-linked immunosorbent assay (ELISA). Same participant may have positive ADA result at more than 1 time point.
Time Frame: pre-dose on Day 1 (Baseline), Week 8, 16, 24, 32
Population: ITT analysis set. Here 'overall number of participants analyzed' signifies participants who were evaluable for this measure at any time point and 'number analyzed' signifies participants who were evaluable at specific time points for each arm, respectively. This outcome was not planned to be analyzed for the 'placebo" arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 71 | 70
Participants
  Baseline: number analyzed (Participants) | 65 | 64
  Baseline | 1 | 2
  Week 8: number analyzed (Participants) | 55 | 55
  Week 8 | 1 | 0
  Week 16: number analyzed (Participants) | 29 | 33
  Week 16 | 0 | 0
  Week 24: number analyzed (Participants) | 55 | 51
  Week 24 | 2 | 0
  Week 32: number analyzed (Participants) | 6 | 8
  Week 32 | 0 | 0

39. Secondary Outcome: Plasma Trough Concentration of Tanezumab
Description: Plasma trough concentration of tanezumab was measured using a validated, sensitive and specific enzyme-linked immunosorbent assay (ELISA).
Time Frame: pre-dose on Day 1 (Baseline), Weeks 8, 16, 24, and 32
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 65 | 65
nanogram per milliliter (ng/mL)
  Baseline | 84.38 (482.59) | 35.68 (176.41)
  Week 8: number analyzed (Participants) | 55 | 54
  Week 8 | 144.2 (95.415) | 342.3 (183.27)
  Week 16: number analyzed (Participants) | 29 | 34
  Week 16 | 188.3 (131.70) | 554.9 (280.30)
  Week 24: number analyzed (Participants) | 55 | 51
  Week 24 | 63.94 (90.513) | 279.5 (422.57)
  Week 32: number analyzed (Participants) | 6 | 8
  Week 32 | 34.15 (53.407) | 95.90 (53.859)

40. Other Pre Specified Outcome: Number of Participants With Intravenous Doses of Study Medication
Description: Number of participants are reported based on the maximum number of intravenous (IV) doses of either tanezumab or placebo received.
Time Frame: Day 1 up to Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
Participants
  1 dose | 41 | 40 | 33
  2 doses | 16 | 16 | 16
  3 doses | 16 | 18 | 23

41. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both serious AEs and non-serious AEs.
Time Frame: Baseline through 112 days after last Intravenous dose of Investigational product to last participant treated with study medication on study (up to Week 32 after last IV dose of investigational product to last participant treated)
Population: as for outcome 40
Measure: Number; unit: participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Number analyzed (Participants) | 73 | 74 | 72
participants
  AEs | 41 | 48 | 39
  SAEs | 0 | 3 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/73 | 3/74 | 0/72
Other Adverse Events (participants affected / at risk) | 36/73 | 39/74 | 29/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 5 mg (N=73) | Tanezumab 10 mg (N=74) | Placebo (N=72)
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 5 mg (N=73) | Tanezumab 10 mg (N=74) | Placebo (N=72)
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0
Oedema peripheral (General disorders) | 3 | 6 | 1
Cellulitis (Infections and infestations) | 0 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 2
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 2
Bacterial test positive (Investigations) | 0 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 15 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 5 | 5
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2
Allodynia (Nervous system disorders) | 0 | 3 | 0
Decreased vibratory sense (Nervous system disorders) | 0 | 0 | 2
Dysaesthesia (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 2
Hyperaesthesia (Nervous system disorders) | 2 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 6 | 4 | 2
Hyporeflexia (Nervous system disorders) | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 12 | 9 | 2
Sciatica (Nervous system disorders) | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Hypertension (Vascular disorders) | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Due to US FDA imposed clinical hold (effective 23 June 2010), study was terminated early and planned sample size was not achieved. Due to change in planned analysis pre-specified outcome measure 'time to discontinuation due to lack of efficacy' was removed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.